CLINICAL TRIAL: NCT03143907
Title: Mindfulness Group-based Intervention for Early Psychosis: A Multi-Site Randomized Control Trial
Brief Title: Mindfulness Group-based Intervention for Early Psychosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: University of Western Ontario, Canada (Other); London Health Sciences Centre (Other); Mindfulness Without Borders (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 108941
Record Dates: First submitted 2017-05-04; First posted 2017-05-08 (Actual); Last update posted 2020-09-24 (Actual); Status verified 2020-09

CONDITIONS: Psychotic Disorders; Schizophrenia
Keywords: Mindfulness; Group Therapy
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia

STUDY DESIGN:
Intervention Model Description: Five sites in total are participating. Three of the five sites are following a RCT design (randomized group allocation; treatment and control group). Two of the five sites are following a pre-post design (no randomized allocation and no control group).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group-A - Immediate Intervention (Other): Immediate Mindfulness Ambassador Council for Early Psychosis (MAC-EP)
  Interventions: Behavioral: Mindfulness Ambassador Council for Early Psychosis (MAC-EP)
- Group-B - Delayed Intervention (Other): 6 month treatment as usual waitlist followed by Mindfulness Ambassador Council for Early Psychosis (MAC-EP)
  Interventions: Behavioral: Mindfulness Ambassador Council for Early Psychosis (MAC-EP)

INTERVENTIONS:
Behavioral: Mindfulness Ambassador Council for Early Psychosis (MAC-EP) — MAC is a 12-week facilitated group mindfulness intervention promoting the development of social-emotional competence in youth created by Mindfulness Without Borders (MWB; www.mwb.org). A meditative practice, mindfulness focuses one's awareness on the present, acknowledging and accepting without judging one's feelings, thoughts, or bodily sensations. Each session has a unique focus (e.g., paying attention, practicing gratitude) and consists of facilitated group learning, discussion and mindfulness skills practice. Home assignments to help reinforce specific lesson are also assigned. MAC has demonstrated acceptability, feasibility, and promising beneficial effects in schools, and in the pilot study conducted at the Early Psychosis Program at London Health Sciences Centre in London, Ontario. Its youth-focus and emphasis on building social and emotional competencies through mindfulness make it a promising intervention for youth recovering from their first episode of psychosis.

SUMMARY:
Recent research has suggested that mindfulness-based interventions (MBI) for psychosis may be effective in reducing the negative symptoms of schizophrenia (e.g., social withdrawal, lack of motivation) and the distress associated with psychotic symptoms (e.g., hearing voices) and could lead to improvements in functioning and quality of life. MBI research to date has primarily focused on studies of patients with chronic psychotic illness, yet relatively little is known about the use of MBIs for youth recovering from their first episode of psychosis. Results from recently published pilot studies appear promising in terms of the feasibility, acceptability, and potential clinical utility (e.g., improved psychological symptoms) of MBIs for the early psychosis population (Ashcroft et al., 2012; van der Valk et al., 2013; Khoury et al., 2015). The current project team has completed a pilot study at the Prevention and Early Intervention Program for Psychoses (PEPP) at London Health Sciences Centre (LHSC), wherein the "Mindfulness Ambassador Council" (MAC), a 12-week facilitated group intervention promoting mindfulness skills and the development of emotional and social competencies, was shown to be an effective, feasible, and acceptable means of treating youth in the early stages of psychotic illnesses. In follow up to the initial pilot study, the purpose of this study is to perform a multi-site Randomized Control Trial to determine the effectiveness of the MAC group intervention on reducing psychotic disorder symptomatology for transitional aged youth experiencing early psychosis. The main hypothesis, based on previous findings on the use of MBIs in psychotic disorders, including results from our initial pilot study at PEPP, is that people with early psychosis who participate in the MAC group intervention will experience improvement in mindfulness skills and affective symptoms compared to those receiving treatment as usual (TAU). Furthermore, we expect that people experiencing early psychosis who participate in MAC will have an improvement in their negative symptoms, quality of life, recovery (self-esteem, perceived recovery), perceived coping, assertiveness, social functioning, and cognitive skills, and a reduction in healthcare service utilization (e.g., emergency room visits, inpatient admissions/length of hospitalization).

DETAILED DESCRIPTION:
The purpose of this multi-site RCT is to determine the effectiveness of the MAC group intervention on reducing psychotic disorder symptomatology (primary outcome) as well as promoting quality of life, critical skills for recovery and decreasing mental health service utilization (secondary outcomes) for transitional aged youth (16-25 years old) experiencing early psychosis. This study is being run at five southern Ontario Early Psychosis Intervention (EPI) sites with Prevention and Early Intervention Program for Psychoses (PEPP) at London Health Sciences Centre (LHSC) being the lead site. Three of the larger sites (located in London, Kitchener-Waterloo, and Hamilton Ontario) are following the RCT design, while the two smaller sites (located in Chatham-Kent and Sarnia, Ontario) are participating in a pre-post design.

For the three RCT sites we aim to recruit 20-24 participants, and for the pre-post sites we aim to recruit 10 participants (total n=92 participants). Participants at the RCT sites will be randomized into Group-A (n = 12; immediate treatment intervention group) or Group-B (n = 12; delayed treatment intervention group). Group-A will receive the MAC intervention at the onset of the study, while Group-B will receive treatment as usual (TAU). Group-B will have the option of receiving the MAC intervention approximately 6 months after the onset of the study. At all times during this study, participants who are receiving the MAC intervention will also be able to continue receiving TAU. Both groups will be assessed with a battery of quantitative measures at baseline (T1), three months later (i.e., immediately post-MAC intervention) (T2), and again three months post-MAC intervention (T3). The measures include interview assessments of psychotic disorder symptoms, and self-report measures of affect, self-esteem, quality of life, coping strategies, assertiveness, social functioning, mindfulness and cognitive skills. In addition, healthcare utilization records for the 6 months preceding MAC intervention onset and for the 6 month duration of the study (3 month MAC intervention + 3 month post-MAC intervention follow-up period) will be collected. Researchers conducting symptom assessment interviews and data analysis will be blinded to the group membership of participants. For the two pre-post sites, all 10 participants will receive the MAC intervention immediately. All 10 participants will complete T1, T2, and T3 assessments and their healthcare utilization records will also be collected.

Based on the pilot study at PEPP-LHSC, and based on previous findings of Mindfulness Based Interventions for psychoses in the literature, we are expecting that participation in the MAC intervention will result in improvement in the following areas: psychotic symptomology (including affective symptoms), mindfulness skills, quality of life, measures of recovery (self-esteem, perceived recovery), perceived coping, assertiveness, social functioning, cognitive skills, and a reduction in healthcare service utilization (e.g., emergency room visits, inpatient admissions/length of hospitalization).

ELIGIBILITY:
Inclusion Criteria:

* Participants must currently be in treatment for psychosis at one of the five Early Psychosis Intervention (EPI) study sites. In addition, participants must have been involved in the program for a period of less than 3 years, due to the focus of this study being on the treatment of early psychosis. Participants must be fluent in English, as determined by referring clinicians or researchers (in the case of advertisement referred participants) in order to meaningfully participate in the MAC intervention and complete the assessment tools.

Exclusion Criteria:

* Potential participants that show high levels of disorganized or disruptive behaviour (as determined by a cut off score of 4 or 5 on the Positive Formal Thought Disorder or Bizarre Behaviour items of the Scale for the Assessment of Positive Symptoms [SAPS]) such that they will not be able to meaningfully participate in the MAC intervention will be excluded from the study.

Ages: 16 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Actual)
Dates: Start 2018-02-22 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Self-Evaluation of Negative Symptoms (SNS) | Baseline, change from Baseline in SNS at 3 months, change from Baseline in SNS at 6 months
  Self-report measure for the assessment of negative symptoms
Kentucky Inventory of Mindfulness Skills | Baseline, change from Baseline in KIMS at 3 months, change from Baseline in KIMS at 6 months
  Self-report measure of mindfulness skills

SECONDARY OUTCOMES:
Rosenberg Self-Esteem Scale (RSES) | Baseline, change from Baseline in RSES at 3 months, change from Baseline in RSES at 6 months
  self-report measure of self-esteem
Profile of Mood States - Short Form (POMS-SF) | Baseline, change from Baseline in POMS-SF at 3 months, change from Baseline in POMS-SF at 6 months
  self-report measure of mood
World Health Organization Quality of Life Scale - Brief version (WHOQOL-BREF) | Baseline, change from Baseline in WHOQOL at 3 months, change from Baseline in WHOQOL at 6 months
  self-report measure of quality of life
Ways of Coping Questionnaire (WCQ) | Baseline, change from Baseline in WCQ at 3 months, change from Baseline in WCQ at 6 months
  self-report measure of ways to cope
Cognitive Failures Questionnaire (CFQ) | Baseline, change from Baseline in CFQ at 3 months, change from Baseline in CFQ at 6 months
  self-report measure of cognitive failures
Rathus Assertiveness Scale (RAS) | Baseline, change from Baseline in RAS at 3 months, change from Baseline in RAS at 6 months
  self-report measure of assertiveness
Health Care Utilization Records Post-Intervention | Utilization at Baseline and during the 6 months following the mindfulness intervention
  form to document participant health care utilization
Kentucky Inventory of Mindfulness Skills (KIMS) | Baseline, change from Baseline in KIMS at 3 months, change from Baseline in KIMS at 6 months
  self-report measure of mindfulness skills
Maryland Assessment of Recovery in People With Serious Mental Illness (MAR) | Baseline, change from Baseline in MAR at 3 months, change from Baseline in MAR at 6 months
  self-report measure of perceived self-recovery
First-Episode Social Functioning Scale (FESFS) | Baseline, change from Baseline in FESFS at 3 months, change from Baseline in FESFS at 6 months
  self-report measure of social functioning

CONTACTS AND LOCATIONS:
Overall Officials: Arlene MacDougall, M.Sc. M.D., Principal Investigator — University of Western Ontario/London Health Sciences Centre
Locations (5):
- Canada (5):
  - Canadian Mental Health Association Chatham-Kent Health Alliance, Chatham, Ontario
  - Canadian Mental Health Association Wellington-Waterloo, Guelph, Ontario
  - Cleghorn Early Psychosis Intervention Clinic, Hamilton, Ontario
  - Prevention and Early Intervention Program for Psychoses, London, Ontario
  - Canadian Mental Health Association Lambton-Kent, Sarnia, Ontario

REFERENCES:
- [Background] Khoury B, Lecomte T, Fortin G, Masse M, Therien P, Bouchard V, Chapleau MA, Paquin K, Hofmann SG. Mindfulness-based therapy: a comprehensive meta-analysis. Clin Psychol Rev. 2013 Aug;33(6):763-71. doi: 10.1016/j.cpr.2013.05.005. Epub 2013 Jun 7. PMID 23796855
- [Background] Khoury B, Sharma M, Rush SE, Fournier C. Mindfulness-based stress reduction for healthy individuals: A meta-analysis. J Psychosom Res. 2015 Jun;78(6):519-28. doi: 10.1016/j.jpsychores.2015.03.009. Epub 2015 Mar 20. PMID 25818837
- [Background] Bell MD, Corbera S, Johannesen JK, Fiszdon JM, Wexler BE. Social cognitive impairments and negative symptoms in schizophrenia: are there subtypes with distinct functional correlates? Schizophr Bull. 2013 Jan;39(1):186-96. doi: 10.1093/schbul/sbr125. Epub 2011 Oct 5. PMID 21976710
- [Background] Birchwood M, Todd P, Jackson C. Early intervention in psychosis. The critical period hypothesis. Br J Psychiatry Suppl. 1998;172(33):53-9. PMID 9764127
- [Background] Shonin E, Van Gordon W, Griffiths MD. Mindfulness-based interventions: towards mindful clinical integration. Front Psychol. 2013 Apr 18;4:194. doi: 10.3389/fpsyg.2013.00194. eCollection 2013. No abstract available. PMID 23616779
- [Background] Shonin E, Van Gordon W, Griffiths MD. Do mindfulness-based therapies have a role in the treatment of psychosis? Aust N Z J Psychiatry. 2014 Feb;48(2):124-7. doi: 10.1177/0004867413512688. Epub 2013 Nov 12. No abstract available. PMID 24220133
- [Background] Norman RM, Manchanda R, Malla AK, Windell D, Harricharan R, Northcott S. Symptom and functional outcomes for a 5 year early intervention program for psychoses. Schizophr Res. 2011 Jul;129(2-3):111-5. doi: 10.1016/j.schres.2011.04.006. Epub 2011 May 5. PMID 21549566
- [Background] Chambers R, Lo BCY, Allen NB. The impact of intensive mindfulness training on attentional control, cognitive style and affect. Cognitive Therapy & Research 32: 303-322, 2008.
- [Background] Buchanan RW. Persistent negative symptoms in schizophrenia: an overview. Schizophr Bull. 2007 Jul;33(4):1013-22. doi: 10.1093/schbul/sbl057. Epub 2006 Nov 10. PMID 17099070
- [Background] Tan LB, Lo BC, Macrae CN. Brief mindfulness meditation improves mental state attribution and empathizing. PLoS One. 2014 Oct 17;9(10):e110510. doi: 10.1371/journal.pone.0110510. eCollection 2014. PMID 25329321
- [Background] Wenk-Sormaz H. Meditation can reduce habitual responding. Altern Ther Health Med. 2005 Mar-Apr;11(2):42-58. PMID 15819448
- [Background] Zeidan F, Johnson SK, Diamond BJ, David Z, Goolkasian P. Mindfulness meditation improves cognition: evidence of brief mental training. Conscious Cogn. 2010 Jun;19(2):597-605. doi: 10.1016/j.concog.2010.03.014. Epub 2010 Apr 3. PMID 20363650
- [Background] Chadwick P, Hughes S, Russell D, Russell I, Dagnan D. Mindfulness groups for distressing voices and paranoia: a replication and randomized feasibility trial. Behav Cogn Psychother. 2009 Jul;37(4):403-12. doi: 10.1017/S1352465809990166. Epub 2009 Jun 23. PMID 19545481
- [Background] Chadwick P, Strauss C, Jones AM, Kingdon D, Ellett L, Dannahy L, Hayward M. Group mindfulness-based intervention for distressing voices: A pragmatic randomised controlled trial. Schizophr Res. 2016 Aug;175(1-3):168-173. doi: 10.1016/j.schres.2016.04.001. Epub 2016 Apr 14. PMID 27146475
- See also: Heinssen, R.K., Goldstein, A.B., & Azrin, S.T. (2014). Evidence-Based Treatments for First Episode Psychosis: Components of Coordinated Specialty Care. Recovery After An Initial Schizophrenia Episode (RA1SE). — http://www.nimh.nih.gov/health/topics/schizophrenia/raise/nimh-white-paper-csc-for-fep_147096.pdf
- See also: Mindfulness Without Borders — http://www.mwb.org